CLINICAL TRIAL: NCT05473078
Title: Attitudes of General Practitioners in Lorraine Towards Prediabetes
Acronym: PréDiabMedG
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, EVA FEIGERLOVA, associate professor, Central Hospital, Nancy, France
Other Study IDs: 2022
Record Dates: First submitted 2022-07-22; First posted 2022-07-25 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: PreDiabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: online anonymous exploratory study — online self-administered questionnary

SUMMARY:
Screening for the risk factors of type 2 diabetes is a part of the primary prevention approach. Pre-diabetes is one of the modifiable risk factors; however, it remains under-diagnosed. Our aim was to analyse the attitudes of general practitioners in Lorraine towards prediabetes

ELIGIBILITY:
Inclusion Criteria:

* General practitioner
* Practice in Lorraine
* Installed or substitute
* Exclusively private practice or mixed activity

Exclusion Criteria:

* Retired physicians
* General practitioners working exclusively in hospital

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: general practitioners
Sampling Method: Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-07-22 (Actual)

PRIMARY OUTCOMES:
Evaluate the attitudes by general practitioners towards pre-diabetes | 4 months
  answers to self-administered questionnary

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: No